CLINICAL TRIAL: NCT01535885
Title: A Phase I Study Of Using Multi-virus Cytotoxic T-cells Following T-cell Depleted Allogeneic Hematopoietic Progenitor Cell Transplantation For Prophylaxis Against Specific Pathogens- Epstein Barr Virus, Adenovirus, And Cytomegalovirus (ACE)
Brief Title: Using Multi-virus Cytotoxic T-cells Following T-Cell Depleted Allogeneic HPCT for Prophylaxis Against EBV, ADV, and CMV
Acronym: ACE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Julie-An M. Talano, Associate Professor of Pediatrics and Director of Clinical Pediatric BMT Research, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CTL-11/157
Record Dates: First submitted 2012-02-06; First posted 2012-02-20 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Epstein-Barr Virus Infections; Adenovirus; Cytomegalovirus Infections
Keywords: Cytoxic T Lymphocytes(CTL); T-cell Depleted; Allogeneic Transplant; Epstein Barr Virus; Adenovirus; Cytomegalovirus; Hematopoietic progenitor cell transplantation
MeSH Terms: conditions — Epstein-Barr Virus Infections; Adenoviridae Infections; Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multi-Virus CTLs (Experimental): The treatment plan delivers a single dose of Multi-Virus CTL to all patients enrolled on study.
  Interventions: Biological: Cytotoxic T Lymphocytes

INTERVENTIONS:
Biological: Cytotoxic T Lymphocytes — Patients will be studied in cohorts of 3. Eligible patients will receive a single Multi-Virus CTL line infusion 28-100 days after their transplant. The dose will start at dose level 1 (2.0 x 106/kg). After each cohort of 3 patients has been treated at each of the dose levels, decisions will be made if the next high or lower dose level should be used.

SUMMARY:
This protocol is a phase I study. Patients may be eligible for an infusion of Multi-virus Cytotoxic T Lymphocytes (CTL) if they received a T-cell depleted (TCD) transplant from a related family member or an unrelated donor. Recipients of these types of transplants are severely immune compromised during the early post-transplant period and are more susceptible to certain viruses. The investigators hypothesize that the adoptive transfer of Cytotoxic T Lymphocytes (CTL) against certain viruses: Adenovirus, Cytomegalovirus and Epstein Barr Virus (Ad, CMV, and EBV) will be safe with regard to producing graft versus host disease (GVHD) or other infusion related toxicities.

DETAILED DESCRIPTION:
Within this clinical trial, the investigators will test the hypotheses that the administration of CTLs for prophylaxis against Ad, CMV and EBV in recipients of TCD-HPCT will be safe and well tolerated. Graded doses of Multi-Virus CTL will be administered to recipients of genotypically haploidentical or mismatched unrelated TCD grafts.

ELIGIBILITY:
Inclusion Criteria:

* Patient age < 22 years.
* Both genders and all races are eligible.
* The patient population chosen for the T-cell depleted allogeneic HPCT from a related or unrelated allogeneic donor must meet eligibility based on institutional SOPs and/or the IRB approved T cell depleted allogeneic HPCT protocol which they are enrolled.
* Must be willing to sign a written informed consent.
* Patient Organ Status at the time of enrollment (pre-transplant)

  * Lansky or Karnofsky score > 50
  * Echocardiogram shortening fraction > 27%
  * Renal function: serum creatinine < 2 x normal for age
  * DLCO > 50% predicted in patients old enough to comply with PFTs or no baseline oxygen requirement for younger patients.
  * Hepatic: AST, ALT < 5x upper limit of normal; bilirubin < 2.0 mg/dl
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months following CTL infusion. The male partner should use a condom.
* Patients must be between 28 and 100 days post T-cell depleted allogeneic HPCT
* Patients must meet the following criteria (within 72 hours of CTL infusion):

  * Achieved primary engraftment with an ANC of at least 1000 per μl for 3 consecutive days.
  * No oxygen requirement with oxygen saturations > 90%.
  * AST, ALT < 5x upper limit of normal for age; bilirubin < 2 mg/dl.
  * Hemoglobin > 8 gm/dl prior to infusion. (May be transfusion dependent).
  * Renal function: serum creatinine < 2 x normal for age.
* The Patient must not have the following conditions on the day of CTL infusion:

  * Exhibit overt hematologic manifestations of relapse or persistent disease.
  * Evidence of recurrent/persistent disease based primarily on flow cytometry, cytogenetics, chimerism analysis, or other molecular studies does not by itself represent grounds for exclusion.

Exclusion Criteria:

* Currently enrolled on another Phase I clinical trial.
* Pregnant or nursing
* Overt hematologic manifestations of relapse or persistent disease
* Having > grade 1 graft-versus-host disease.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
To assess toxicity by SAEs scored according to the adaptive CTCAE version 5 | 1 year
  Phase/safety/toxicity

SECONDARY OUTCOMES:
Evidence of immunity against specific viral pathogens- Ad, CMV and EBV in recipients of Multi-Virus CTLs | 1 year
  Immunity will be recorded.
The incidence of Ad, EBV, and CMV systemic infections during the first 180 days post-transplant | 1 year
  Number of infections will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Julie-An Talano, MD, Principal Investigator — Medical College of Wisconsin/Children's Hospital of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States